CLINICAL TRIAL: NCT05824559
Title: A Phase 1b Study of the OxPhos Inhibitor ME-344 Combined With Bevacizumab in Previously Treated Metastatic Colorectal Cancer
Brief Title: ME-344 and Bevacizumab in Previously Treated Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision to wind down operations, close all clinical programs and evaluate strategic options
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-344-003
Record Dates: First submitted 2023-03-22; First posted 2023-04-21 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ME-344; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b open-label, multiple dose/schedule sequential study to determine the safety and efficacy of the oxidative phosphorylation (OxPhos) pathway inhibitor ME-344 in combination with bevacizumab in subjects with recurrent mCRC.
  Subjects in Cohort 1 will receive ME-344 (IV) on Days 1, 8 and 15 combined with bevacizumab (IV) on Days 1 and 15 of each 28-day cycle.
  Subjects in Cohort 2 will receive ME 344 (IV) on Days 1 and 15 combined with bevacizumab (IV) on Days 1 and 15 of each 28-day cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ME-344 and Bevacizumab (Experimental): ME-344 (IV) Cohort 1: Days 1, 8, and 15 of each 28-day cycle. Cohort 2: Days 1 and 15 of each 28-day cycle.
  Bevacizumab (IV) Cohorts 1 and 2: Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: ME-344; Drug: Bevacizumab

INTERVENTIONS:
Drug: ME-344 — ME-344 will be administered intravenously (IV)
Drug: Bevacizumab — Bevacizumab will be administered intravenously (IV)

SUMMARY:
This is a Phase 1b open-label, multiple dose/schedule sequential study to determine the safety and efficacy of the oxidative phosphorylation (OxPhos) pathway inhibitor ME-344 in combination with bevacizumab in subjects with recurrent mCRC.

DETAILED DESCRIPTION:
This is a Phase 1b open-label, multiple dose/schedule sequential study to determine the safety and efficacy of the oxidative phosphorylation (OxPhos) pathway inhibitor ME-344 in combination with bevacizumab in subjects with recurrent mCRC.

This study will enroll subjects with metastatic CRC, including but not limited to subjects with RAS wild-type or mutant tumors, MSI-H/pMMR, and BRAF V600E, who have progressed or demonstrated intolerability to standard approved therapies which include fluoropyrimidine, oxaliplatin, irinotecan-based chemotherapies, cetuximab/panitumumab, PD-1 inhibitors, or BRAF inhibitors (if clinically indicated), and/or other checkpoint inhibitors. Approximately 40 subjects will be enrolled in the study, in 2 cohorts of 20 subjects each.

Subjects will continue treatment with ME-344 and bevacizumab until radiological progressive disease, unacceptable AEs, withdrawal of consent, start of new anticancer therapy, or death.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histological or cytological documentation of adenocarcinoma of the colon or rectum that is metastatic (all other histological types are excluded)
* Subjects who progressed or demonstrated intolerability to prior standard approved therapies which include fluoropyrimidine, oxaliplatin, and irinotecan-based chemotherapies, cetuximab/panitumumab (if clinically indicated e.g., RAS wild-type tumors) PD-1 or BRAF inhibitors (if clinically indicated), and/or other checkpoint inhibitors in the metastatic setting.
* Previous treatment with any investigational drug or anticancer treatment must be completed >28 days or 5 half-lives, whichever is longer, before the first dose of study treatment.
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Untreated brain metastases, spinal cord compression, or primary brain tumor
* Symptomatic brain metastases, leptomeningeal disease, spinal cord compression, or primary brain tumor
* Evidence of uncontrolled or unstable cardiovascular disease, myocardial infarction (within 6 months), unstable angina pectoris, congestive heart failure, serious arrhythmias requiring drug therapy
* History of CNS disease
* Bevacizumab or aflibercept therapy ≤ 3 weeks prior to starting study treatment
* Peripheral neuropathy Grade ≥ 2
* Uncontrolled hypertension or diabetes mellitus, active peptic ulcers, unhealed wounds, clinically significant disease or systemic infections
* Known seropositive for, or active infection with hepatitis B or C virus
* Symptomatic or uncontrolled infection with human T-cell leukemia virus
* Venous thromboembolism (unless appropriately treated and stable on anticoagulant for at least 2 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California, Los Angeles, California
  - Mount Sinai Miami, Miami Beach, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Rutgers University, New Brunswick, New Jersey
  - Mt Sinai New York, New York, New York
  - Vanderbilt -Ingram Cancer Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Boland PM, Lenz HJ, Ciombor KK, Florou V, Pishvaian MJ, Cusnir M, Cohen D, Guo JY, Tang M, Rajagopalan P, Wiley SE, Ghalie RG, Hochster HS. A Phase 1b study of the OxPhos inhibitor ME-344 with bevacizumab in refractory metastatic colorectal cancer. Invest New Drugs. 2025 Feb;43(1):60-68. doi: 10.1007/s10637-024-01489-1. Epub 2024 Dec 27. PMID 39725778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open from August of 2023 to July 2024 at 7 centers in the United States. 23 subjects were enrolled. Due to business reasons this study was terminated in July of 2024, and Cohort 2 was never opened.
Groups:
- ME-344 and Bevacizumab: ME-344 10 mg/kg (IV) Cohort 1: given on Days 1, 8, and 15 of each 28-day cycle.
  Bevacizumab 5 mg/kg IV Cohort 1: given on Days 1 and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | ME-344 and Bevacizumab
Started | 23
Completed | 0
Not Completed | 23
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Progressive Disease | 16
Not completed — Study Terminated by Sponsor | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | ME-344 and Bevacizumab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at 16 Weeks
Description: Progression Free Survival is measured by using laboratory testing and scans. It is measured by the length of time from first dose of study drug until observation of disease progression.
Time Frame: 16 weeks
Population: All patients had relapsed metastatic colorectal cancer.
Measure: Number; unit: percentage
Arm/Group | ME-344 and Bevacizumab
Number analyzed (Participants) | 23
percentage | 31.8

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) is defined/measured by the proportion of patients achieving complete response [CR] or partial response [PR] per RECIST v.1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ME-344 and Bevacizumab
Number analyzed (Participants) | 23
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 9
  Progressive Disease | 10
  Not Available | 4

3. Secondary Outcome: Treatment Emergent Adverse Events for ME-344 Administered in Combination With Bevacizumab
Description: This will be measured by the number of participants with at least one treatment emergent Adverse Events (abnormal physical examination findings, abnormal vital signs, abnormal ECG QT interval and abnormal clinical laboratory results)
Time Frame: from first dose of study drug on Cycle 1 Day 1 through 30 days after the last dose of study drug or start of new anticancer treatment, up to 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | ME-344 and Bevacizumab
Number analyzed (Participants) | 23
Participants | 22

ADVERSE EVENTS:
Time Frame: from first dose of study drug on Cycle 1 Day 1 through 30 days after the last dose of study drug or start of new anticancer treatment, up to 11 months
Arm/Group | ME-344 and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ME-344 and Bevacizumab (N=23)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ME-344 and Bevacizumab (N=23)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 11 (11)
Non-cardiac chest pain (General disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Prostate infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 (1)
Stoma obstruction (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood sodium decreased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (3)
Blood albumin decreased (Investigations) | 2 (2)
Blood potassium decreased (Investigations) | 2 (2)
Urine protein/creatinine ratio increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Blood calcium increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Urine potassium increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Anorexia nervosa (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT05824559/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT05824559/SAP_001.pdf